CLINICAL TRIAL: NCT03906214
Title: Evidence-based Assessment of Medication Sensitivity in Acute Hepatic Porphyria
Status: Completed | Type: Observational
Sponsor: University of South Florida (Other)
Collaborators: University of Texas (Other); Wake Forest University Health Sciences (Other); University of Miami (Other); University of Washington (Other); Icahn School of Medicine at Mount Sinai (Other); University of Alabama at Birmingham (Other); University of California, San Francisco (Other); University of Utah (Other); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Other Study IDs: PC 7208
Record Dates: First submitted 2019-04-04; First posted 2019-04-08 (Actual); Last update posted 2019-10-16 (Actual); Status verified 2019-04

CONDITIONS: Porphyrias
Keywords: Porphyrias; Variegate Porphyria; Hereditary Coproporphyria; Acute Intermittent Porphyria
MeSH Terms: conditions — Porphyrias; Porphyria, Variegate; Coproporphyria, Hereditary; Porphyria, Acute Intermittent

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Web-based Survey — Participants will be directed to online forms to report general information (ex. age, sex, test results, family history), suspected medication-related acute attacks, and "uneventful use of possibly risky medication". If a patient has multiple medication-related acute attacks, the patient/caregiver will be able to submit multiple report forms that will be linked. In addition to the report forms, patients will be asked to review a list of "Medications of Interest" and report current or past use.

SUMMARY:
This is an observational study collecting patient/caregiver reports on suspected medication/drug-induced acute porphyria attacks, as well as safe use of drugs previously labeled "unsafe" or with unknown risk. Participants will be recruited through the RDCRN Contact Registry for the Porphyrias Consortium. The study will be advertised on the Consortium website and through the American Porphyria Foundation's social media network.

DETAILED DESCRIPTION:
Contact Registrants will be sent an email invitation describing the study. A unique link will be generated for each registrant and included in the email invitation. After 2 weeks, a second email invitation will be sent to the registrants who have not yet participated. After 1 month, a third email invitation will be sent to the registrants who have not yet participated. We may send additional emails periodically (e.g. every 6-12 months) to subjects enrolled to remind them to complete new surveys if they have taken any other medications of interest or have experienced any new reactions/attacks.

If the registrant wants to participate in the study, he/she will follow the survey link in the email invitation, which directs him/her to an IRB-approved online consent form. If the participant consents to participate, he/she will be directed to online forms to report general information (ex. age, sex, test results, family history), suspected medication-related acute attacks, and "uneventful use of possibly risky medication". If a patient has multiple medication-related acute attacks, the patient/caregiver will be able to submit multiple report forms that will be linked. In addition to the report forms, patients will be asked to review a list of "Medications of Interest" and report current or past use.

ELIGIBILITY:
Inclusion Criteria:

* Able to read and write in English
* Enrolled in the RDCRN PC Contact Registry
* Self-reported patient or caregiver of patient with acute porphyria

There are no restrictions on age, sex or ethnicity. However, the following criteria will be applied to those reports that are considered evaluable (analyzed and scored):

1. Medication name must be specified
2. The data elements required in the scoring system must be complete

Exclusion Criteria:

* Unable to provide informed consent and complete forms

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants will be recruited through the RDCRN Contact Registry for the Porphyrias Consortium.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2019-04-03 (Actual); Primary Completion 2019-09-13 (Actual); Study Completion 2019-09-13 (Actual)

PRIMARY OUTCOMES:
Acute Attack Form | 5 years from study start
  Designed to capture PBG levels, characteristics of the acute attack, timing of medication administration, and pharmacological information on the medication.
Uneventful Use of Possible Risky Medication Form | 5 years from study start
  Designed to capture details of medication in question, ALA/PGB results during use of medication in questions, concomitant medication use, diet history, and alcohol use.
Use of Medications of Interest Form | 5 years from study start
  Designed to assess medications used by category and effects of each.

CONTACTS AND LOCATIONS:
Overall Officials: D. Montgomery Bissell, MD, Study Chair — University of California, San Francisco; Bruce Wang, MD, Study Chair — University of California, San Francisco
Locations (1):
- University of South Florida Data Management Coordinating Center, Tampa, Florida, United States

REFERENCES:
- [Background] Anderson KE, Bloomer JR, Bonkovsky HL, Kushner JP, Pierach CA, Pimstone NR, Desnick RJ. Recommendations for the diagnosis and treatment of the acute porphyrias. Ann Intern Med. 2005 Mar 15;142(6):439-50. doi: 10.7326/0003-4819-142-6-200503150-00010. PMID 15767622
- [Background] de Matteis F. Disturbances of liver porphyrin metabolism caused by drugs. Pharmacol Rev. 1967 Dec;19(4):523-57. No abstract available. PMID 4868613
- [Background] Seth AK, Badminton MN, Mirza D, Russell S, Elias E. Liver transplantation for porphyria: who, when, and how? Liver Transpl. 2007 Sep;13(9):1219-27. doi: 10.1002/lt.21261. PMID 17763398
- [Background] Slavin SA, Christoforides C. Thiopental administration in acute intermittent porphyria without adverse effect. Anesthesiology. 1976 Jan;44(1):77-9. doi: 10.1097/00000542-197601000-00021. No abstract available. PMID 1244784
- [Background] Thunell S, Pomp E, Brun A. Guide to drug porphyrogenicity prediction and drug prescription in the acute porphyrias. Br J Clin Pharmacol. 2007 Nov;64(5):668-79. doi: 10.1111/j.0306-5251.2007.02955.x. Epub 2007 Jun 19. PMID 17578481